CLINICAL TRIAL: NCT00585117
Title: Pilot Study of (61)CuATSM-PET Imaging in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in imaging priorities
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC 2006-0282; RO06309 (Other: UW Carbone Cancer Center); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison)
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2012-02

CONDITIONS: CNS Brain Metastases; Head and Neck Cancer; Lung Cancer; Prostate Cancer; Esophageal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms | interventions — Magnetic Resonance Spectroscopy; CuATSM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 CNS (Experimental): imaging with CuATSM
  Interventions: Procedure: PET-imaging with CuATSM; Procedure: PET Imaging
- 2. Head and Neck (Experimental): Imaging with CuATSM
  Interventions: Procedure: PET CuATSM
- 3. Lung (Experimental): imaging with CuATSM
  Interventions: Procedure: PET imaging
- 4. Prostate (Experimental): PET imaging with CuATSM
  Interventions: Procedure: PET imaging with CuATSM
- 5. Esophagus (Experimental): PET imaging with CuATSM
  Interventions: Procedure: PET imaging with CuATSM

INTERVENTIONS:
Procedure: PET-imaging with CuATSM — imaging with CuATSM
  Arms: 1 CNS
Procedure: PET Imaging — Imaging with CuATSM
  Arms: 1 CNS
Procedure: PET CuATSM — Imaging with CuATSM
  Arms: 2. Head and Neck
Procedure: PET imaging — imaging with CuATSM
  Arms: 3. Lung
Procedure: PET imaging with CuATSM — Imaging with CuATSM
  Arms: 4. Prostate
Procedure: PET imaging with CuATSM — Imaging with CuATSM
  Arms: 5. Esophagus

SUMMARY:
Hypoxia is a key factor in malignant progression of a neoplasm. It is our aim to explore the basis for quantitative in vivo tumor imaging by Cu-61 diacetyl-bis(N4-methylthiosemicarbazone)PET imaging as a surrogate of tissue hypoxia. We hypothesize that the hypoxia levels are predictive of the tumor response to therapy. Patients will have 2 CU-ATSM PET scans done and the goal is to show spatially stable tracer distributions that correlate with tumor hypoxia. This study will serve as a pilot study for a PO1 submission

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerated a PET/CT scan
* Age 18 or older
* Patient being considered for XRT for treatment of their cancer
* Able to provide written informed consent

Exclusion Criteria:

* severe claustrophobia or inability to tolerate the PET scan
* pregnant or breastfeeding women
* Patients that need supplemental oxygen
* Patients enrolled in experimental treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To validate the CuATSM-PET imaging by correlation to the serum level of osteopontin, a marker of hypoxia | end of study

SECONDARY OUTCOMES:
To test reliability of the CuATSM uptake by quantifying the reproducibility of the pre-treatment CuATSM_PET scans | end of study
To assess the technical and logistic feasibility of CuATSM-PET scans in a population of cancer patients | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jeraj, Ph.D, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States